CLINICAL TRIAL: NCT00124995
Title: Double-blinded Randomized Trial of Terbutaline to Shorten ICU Length of Stay in the Treatment of Status Asthmaticus in Children
Brief Title: Trial of Terbutaline for the Treatment of Status Asthmaticus in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Carroll, MD, Associate Professor of Pediatrics, Connecticut Children's Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 05-001
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Status Asthmaticus
MeSH Terms: conditions — Status Asthmaticus | interventions — Terbutaline

INTERVENTIONS:
Drug: terbutaline

SUMMARY:
Although widely used for the treatment of pediatric status asthmaticus, intravenous terbutaline has potentially significant side effects; may not improve outcomes; and may increase Intensive Care Unit (ICU) length of stay. This study is designed to test the efficacy of intravenous terbutaline for the treatment of status asthmaticus by adding intravenous terbutaline or placebo to standard asthma treatment. The dose of terbutaline or placebo will be titrated according to severity of illness as quantified by a validated clinical asthma score. Differences in outcomes between the study groups, such as length of stay, hospital costs, and lung function will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Connecticut Children's Medical Center (CCMC) Pediatric Intensive Care Unit (PICU) with a primary admission diagnosis of status asthmaticus
* Modified Pulmonary Index Score (MPIS) of greater than or equal to 12
* Age between birth and 18 years old

Exclusion Criteria:

* Pre-existing cardiac or pulmonary disease
* Existing respiratory failure (requiring invasive or non-invasive mechanical ventilation)
* Hemodynamic or cardiovascular instability requiring inotropic support
* The patient meets one of the criteria for withdrawal from the study due to patient safety concerns

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2003-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
ICU length of stay

SECONDARY OUTCOMES:
To evaluate the effects of intravenous terbutaline on pulmonary mechanics over length of ICU admission
To prospectively analyze the side effects of terbutaline

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Carroll, MD, Principal Investigator — CT Children's Medical Center
Locations (1):
- CT Children's Medical Center, Hartford, Connecticut, United States